CLINICAL TRIAL: NCT06909708
Title: SIRT (Yttrium-90 Carbon Microspheres) Versus cTACE for Unresectable Hepatocellular Carcinoma: A Multicenter, Prospective, Open-label, Phase 3 Trial (CHANCE2506)
Brief Title: SIRT Versus cTACE for Unresectable HCC (CHANCE2506)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Director of Interventional and Vascular Surgery Department, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHANCE2506-NRT6003
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: HCC; TACE; Selective internal radiation therapy; Yttrium-90
MeSH Terms: interventions — Sirtuins; Yttrium-90

STUDY DESIGN:
Intervention Model Description: Experimental Group : Yttrium-90 carbon microspheres. Control Group : Conventional transarterial chemoembolization (cTACE) using anti-tumor drug, lipiodol and embolic particles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIRT Group (Experimental): Each Participant will underwent a single intra-arterial infusion of yttrium-90 carbon microspheres (NRT6003 injection)].
  Interventions: Procedure: SIRT
- cTACE Group (Active Comparator): Each Participant will underwent conventional transarterial chemoembolization (cTACE).
  Interventions: Procedure: cTACE

INTERVENTIONS:
Procedure: SIRT — Y-90 administered
  Other Names: Yttrium-90 [90Y]
  Arms: SIRT Group
Procedure: cTACE — cTACE administered
  Arms: cTACE Group

SUMMARY:
To evaluate the efficacy and safety of yttrium-90 carbon microspheres versus cTACE in patients with unresectable hepatocellular carcinoma

DETAILED DESCRIPTION:
The efficacy and safety of yttrium-90 carbon microspheres versus in patients with unresectable hepatocellular carcinoma (HCC) remain unknown. This multicenter, prospective, open-label, phase 3 trial is designed to evaluate the safety and efficacy of yttrium-90 carbon microspheres versus conventional TACE in patients with hepatocellular carcinoma. The primary endpoint is time to progression for patients with HCC. While the secondary endpoints include the overall response rate, duration of response, local time to progression, tumor biomarkers variation, overall survival and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group performance status ≤ 1;
2. Expected survival time ≥ 3 months;
3. Confirmed hepatocellular carcinoma based on CNLC guidelines;
4. Without extrahepatic metastases, unresectable or refuse surgical resection;
5. At least one well defined tumor (mRECIST 1.1);
6. Tumor burden≤50% of the total liver volume;
7. Child-Pugh score≤7;
8. Adequate organ function: # Blood routine: absolute neutrophil count ≥ 1.5×10^9/L; platelet≥75×10^9/L; hemoglobin≥90 g/L; # Liver function: total bilirubin≤2 times upper limit of normal (ULN); alanine transaminase and aspartate aminotransferase≤5.0 ULN; alkaline phosphatase≤2.5 ULN; Albumin>30 g/L; # Renal function: Cr≤1.5 ULN; creatinine clearance≥50 mL/min; # Coagulation function: international normalized ratio, prothrombin time and activated partial thromboplastin time were less than 1.5 ULN;
9. Women and men of childbearing age must agree to take strict and effective contraceptive measures during the study period and within 6 m after the end of the trial.

Exclusion Criteria:

1. With previous history of hepatic encephalopathy;
2. Extrahepatic disease or combined with other malignant tumors;
3. Infiltrative hepatocellular carcinoma ;
4. With prior antitumor therapies, including liver transplantation, hepatectomy, ablation, TACE, chemotherapy, radiotherapy, targeted therapy or immunotherapy;
5. With hepatic artery malformation and unable to undergo TACE or SIRT;
6. Allergy to contrast agents or anesthetics
7. With clinical manifestations of portal hypertension, moderate-severe or refractory ascites, or decompensated liver cirrhosis, or moderate-to-severe esophageal/gastric varices;
8. With severe pulmonary insufficiency (forced expiratory volume at one second / forced vital capacity<50% or forced expiratory volume at one second /predicting value<50% or maximum volume per minute<50 L/min);
9. The single lung radiation absorbed dose>30 Gy;
10. Tumor thrombus in main portal vein or hepatic artery or hepatic vein or bile duct;
11. Serious infections in active stage or need systematic treatment;
12. Pregnant and lactating women;
13. With positive results of HIV antibody test;
14. HBV DNA or HCV RNA positive;
15. With active syphilis or tuberculosis;
16. 99mTc-MAA imaging (patients exclusion meet all criteria):

1) Perfusion area covers all intrahepatic tumors (including non-target lesions) and non-perfused liver volume ≥30% of total liver volume; 2) Tumor dose ≥400 Gy for 1-2 hepatic segments; Perfused normal liver dose (PNLD): 120 Gy < PNLD <1000 Gy; Tumor dose ≥200 Gy (recommended ≥400 Gy) and PNLD <120 Gy with other condition; 3) No gastrointestinal shunt , or shunt amendment by endovascular techniques (reassessment required); 4) cTACE should cover all intrahepatic lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | From enrollment to 54 weeks after the treatment
  Evaluated by the independent image review committee (CTCAE 5.0)

SECONDARY OUTCOMES:
Adverse events | From enrollment to 54 weeks after the treatment
  Rates and degree of adverse events
Severe adverse events | From the enrollment to 54 weeks after the treatment.
  Rates of severe adverse events
localized time to progression | From the enrollment to 54 weeks after the treatment.
  Localized time to progression evaluated by the investigator
Objective response rates (ORR) | From enrollment to 54 weeks after the treatment.
  Evaluated by the investigator
Overall survival (OS) | From the enrollment to the death or lost to follow up.
  Overall survival
Duration of response (DoR) | From the enrollment to 54 weeks after the treatment
  Evaluated by the investigator
Resection rate of liver target lesions | From enrollment to 54 weeks after the treatment.
  Resection rate of liver target lesions
Tumor markers | From the enrollment to 54 weeks after the treatment.
  The variation of tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, Principal Investigator — Zhongda Hospital, Soueast University
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No